CLINICAL TRIAL: NCT00360607
Title: A Randomized, Open Label, Multicentre Phase Iv Study To Evaluate The Efficacy And Safety Of Magnex (Cefoperazone-Sulbactam) In Comparison With Ceftazidime Plus Amikacin And Metronidazole In The Treatment Of Intra-Abdominal Infections
Brief Title: A Comparative Phase IV Study Evaluating Efficacy & Safety Of Magnex(Cefoperazone-Sulbactam) In Intraabdominal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1891002
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Sulbactam; Cefoperazone; Ceftazidime; Metronidazole; Amikacin

INTERVENTIONS:
Drug: Magnex (Sulbactam Sodium/Cefoperazone Sodium 1:1) Pfizer Ltd.
Drug: Fortum (Ceftazidime for injection USP) Glaxo Smith Kline Pharmaceuticals Limited
Drug: Metrogyl (Metronidazole Injection IP) J.B.Chemicals & Pharmaceuticals Ltd.
Drug: Mikacin (Amikacin Sulphate Injection IP) Aristo Pharmaceuticals Ltd.

SUMMARY:
Intra-abdominal infections are often polymicrobial, and include aerobic as well as anaerobic bacteria. Antibiotics used in intra-abdominal infections should aim to cover organisms such as Enterobacteriaceae and Bacteroides fragilis, which are the commonest organisms known to cause such infections. Combinations of a third-generation cephalosporin, an aminoglycoside and metronidazole are often used to treat such infections in surgical settings. An alternative to such combinations is the use of a beta lactam - beta lactamase inhibitor combination. Magnex (cefoperazone- sulbactam) is one such combination, which has been shown to be as effective as a standard multidrug regimen such as gentamicin and clindamycin in the management of intra-abdominal infections. The combination of ceftazidime, amikacin and metronidazole has been chosen as a comparator regimen because of its broad coverage of Gram-negative and anaerobic organisms found in such conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged greater or equal to 12 years
* Intra-abdominal infection documented by laparotomy or laparoscopy or percutaneous aspiration within 24 hours prior to screening
* Presence of at least three of the following five indicators consistent with intra-abdominal infections (Fever, leucocytosis, abdominal symptoms, abdominal signs, radiological evaluation)
* Written informed consent obtained

Exclusion Criteria:

* Rapidly progressive illness or critically ill subjects
* Pregnant or lactating women, or women of childbearing potential not using an effective method of contraception.
* Treatment with a presumably effective systemic antimicrobial agent for >24 hours within a 72 hour period prior to study entry unless the subject did not sufficiently respond to the treatment (as judged by the investigator)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2004-07; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Proportion of clinical efficacy-evaluable subjects who present with continued resolution at the 30-day follow-up visit.
Adverse events as observed by the investigator or volunteered as responses to unsolicited and non-leading questions.
Vital signs including systolic and diastolic blood pressures, pulse rate and respiratory rate.
Physical examination findings.

SECONDARY OUTCOMES:
The proportion of clinical efficacy
evaluable subjects who are classified as having a clinical outcome of success or improvement at the end of study treatment;
proportion of microbiological efficacy-evaluable subjects who have a successful microbiological outcome
success or presumed success) at the end of study treatment,
Total duration of study treatment
Comparison of pharmaco-economic data (cost effectiveness) for cefoperazone- sulbactam versus the combination of ceftazidime - amikacin - metronidazole.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- India (16):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Bhopal, Madhya Pradesh
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, Chandigarh
  - Pfizer Investigational Site, Coimbatore
  - Pfizer Investigational Site, Hyderabad
  - Pfizer Investigational Site, Lucknow
  - Pfizer Investigational Site, Ludhiana
  - Pfizer Investigational Site, Mumbai

REFERENCES:
- [Derived] Chandra A, Dhar P, Dharap S, Goel A, Gupta R, Hardikar JV, Kapoor VK, Mathur AK, Modi P, Narwaria M, Ramesh MK, Ramesh H, Sastry RA, Shah S, Virk S, Sudheer OV, Sreevathsa MR, Varshney S, Kochhar P, Somasundaram S, Desai C, Schou M. Cefoperazone-sulbactam for treatment of intra-abdominal infections: results from a randomized, parallel group study in India. Surg Infect (Larchmt). 2008 Jun;9(3):367-76. doi: 10.1089/sur.2007.013. PMID 18570578
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1891002&StudyName=A+Comparative+Phase+IV+Study+Evaluating+Efficacy+%26+Safety+Of+Magnex%28Cefoperazone%2DSulbactam%29+In+Intraabdominal+Infections